CLINICAL TRIAL: NCT01691716
Title: A Prospective Randomized Study Comparing the Therapeutic Effect of Tendoactive®, Eccentric Training, and a Combination of Both as a Treatment of Achilles Tendinopathy
Brief Title: The Efficacy of Tendoactive, Eccentric Training, and the Combination of Both as a Treatment of Achilles Tendinopathy
Acronym: Tendoactive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioiberica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRJ-00014
Record Dates: First submitted 2012-09-13; First posted 2012-09-25 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Achilles Tendinopathy
Keywords: Achilles tendinopathy; Tendoactive; Eccentric training

ARMS (3):
- Tendoactive (Experimental): Tendoactive dosage: 3 capsules per day
  Interventions: Drug: Tendoactive
- Eccentric training (Active Comparator): Protocol published by Alfredson et al 1998 (Am J Sports Med 1998 26: 360)
  Interventions: Behavioral: Eccentric training
- Tendoactive and eccentric training (Active Comparator): Tendoactive dosage: 3 capsules per day. Eccentric training: protocol described by Alfredson et al 1998 (Am J Sports Med 1998 26: 360)
  Interventions: Drug: Tendoactive; Behavioral: Eccentric training

INTERVENTIONS:
Drug: Tendoactive — Food supplement containing mucopolysaccharides, type I collagen and vitamin C
  Arms: Tendoactive; Tendoactive and eccentric training
Behavioral: Eccentric training — Eccentric training program published by Alfredson et al 1998 (Am J Sports Med 1998 26: 360)
  Arms: Eccentric training; Tendoactive and eccentric training

SUMMARY:
The purpose of this study is to determine whether Tendoactive, eccentric training, or the combination or both could be effective in the treatment of Achilles tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from a gradually evolving painful condition in the Achilles tendon located at the midportion for at least 3 months (Diagnosis based on clinical examination showing a painful thickening of the Achilles tendon located at a level of 2 to 6cm above the tendon insertion, and confirmed by ultrasonography: local thickening of the tendon, irregular tendon structure with hypoechoic areas and irregular fiber orientation).
* Men and non-pregnant women aged 18-70 years
* Be informed of the nature of the study and provide written informed consent.

Exclusion Criteria:

* Clinical suspicion of insertional disorders (pain at the site of the insertion of the Achilles tendon on the calcaneum)
* Clinical suspicion of an Achilles tendon rupture (Thompson test abnormal and palpable "gap")
* Clinical suspicion of plantar flexor tenosynovitis (posteromedial pain when the toes are plantar flexed against resistance)
* Clinical suspicion of n.suralis pathology (sensitive disorder in the area of the sural nerve)
* Clinical suspicion of peroneal subluxation
* Suspicion of internal disorders: spondylarthropathy, gout, hyperlipidemia, Rheumatoid Arthritis and sarcoidosis.
* Condition that prevents the patients from executing an active exercise programme
* Patient has already performed eccentric exercises, according to the schedule of Alfredson et al (12 weeks)
* Patient has already received an injection of PRP for this injury
* Patient does not wish, for whatever reason, to undergo one of the two treatments
* Known presence of a pregnancy
* Condition of the Achilles tendon caused by medications (arising in relation to moment of intake), such as quinolones and statins

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in VISA-A score at 12 weeks | 12 weeks
  Functional impairment of the Achilles tendon is measured using VISA-A score. Score of patient-related outcome measure: Achilles tendon: VISA-A [0=worse, 100=perfect] derived from eight validated questions on pain and function during activities of daily living

SECONDARY OUTCOMES:
Pain level at rest [VAS 0-10] | 0, 6, 12 weeks
Pain level at exertion [VAS 0-10] | 0, 6, 12weeks
Achilles transverse thickness by ultrasound | 0, 6, 12 weeks
  Ultrasound evaluation of Achilles tendon. Maximum thickness will be recorded in the midportion of the affected Achilles tendon
SF-36 v2 quality of life survey | 0, 12 weeks
Patient satisfaction | 6, 12 weeks
  Patient satisfaction will be evaluated using a subjective questionnaire.

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - CMI, Barcelona, Barcelona
  - CEARE, Esplugues de Llobregat, Barcelona
  - Clínica CEMTRO, Madrid, Madrid
  - AMS - Centro de Ejercicio, Málaga, Malaga
  - Centro de Medicina y Deporte, Toledo, Toledo
  - Clínica Traumatológica, Valladolid, Valladolid

REFERENCES:
- [Background] Alfredson H, Pietila T, Jonsson P, Lorentzon R. Heavy-load eccentric calf muscle training for the treatment of chronic Achilles tendinosis. Am J Sports Med. 1998 May-Jun;26(3):360-6. doi: 10.1177/03635465980260030301. PMID 9617396
- [Derived] Balius R, Alvarez G, Baro F, Jimenez F, Pedret C, Costa E, Martinez-Puig D. A 3-Arm Randomized Trial for Achilles Tendinopathy: Eccentric Training, Eccentric Training Plus a Dietary Supplement Containing Mucopolysaccharides, or Passive Stretching Plus a Dietary Supplement Containing Mucopolysaccharides. Curr Ther Res Clin Exp. 2016 Nov 18;78:1-7. doi: 10.1016/j.curtheres.2016.11.001. eCollection 2016. PMID 28053674